CLINICAL TRIAL: NCT02557737
Title: Comparison of Surface Landmark, Ultrasonography and Electric Stimulation Guidance for Botulinum Toxin Injections in Stroke Patients With Spasticity on Upper Extremities.
Brief Title: Botulinim Toxin Type A Injections by Different Guidance in Stroke Patients With Spasticity on Upper Extremities
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMRPG8B0222
Record Dates: First submitted 2015-09-17; First posted 2015-09-23 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Cerebrovascular Accident
Keywords: stroke; upper extremity; spasticity; botulinum toxin; ultrasonography; electric stimulation
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — Botulinum Toxins, Type A; Botulinum Toxins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ultrasonography direct-guidance (Experimental): To inject Botulinum toxin type A on the spasticity lower extremity for stroke patients by Ultrasonography direct-guidance.
  Interventions: Drug: Botulinum Toxin Type A
- Electric stimulation (Experimental): To inject Botulinum toxin type A on the spasticity lower extremity for stroke patients by Electric stimulation
  Interventions: Drug: Botulinum Toxin Type A
- Surface anatomy landmark (Active Comparator): To inject Botulinum toxin type A on the spasticity lower extremity for stroke patients by Surface anatomy landmark.
  Interventions: Drug: Botulinum Toxin Type A

INTERVENTIONS:
Drug: Botulinum Toxin Type A — To inject Botulinum toxin type A on the spasticity lower extremity for stroke patients by Ultrasonography direct-guidance, Ultrasonography direct-guidance, Electric stimulation and Surface anatomy landmark.
  Other Names: Botulinum toxin

SUMMARY:
The aims of this study were to compare the injection locations of key spastic muscles on upper extremity by three different guidance localization methods ( surface anatomy landmark, ultrasonography, electric stimulation) and the effectiveness.

DETAILED DESCRIPTION:
Stroke may result in acute or chronic hemiplegia and spasticity in stroke patients. Spasticity in upper extremities may interfere with motor voluntary function, activities of daily living and cause muscle pain. Botulinum toxin type A (BTX-A) has been shown to relieve spasticity and pain in upper extremities of stroke patients. There are no researches to compare the efficiency of BTX-A by different injection guidance methods in stroke patients. The aims of our study were to compare the injection locations of key spastic muscles on upper extremity by three different guidance localization methods ( surface anatomy landmark, ultrasonography, electric stimulation) and the effectiveness. The investigators will enroll 60 hemiplegic stroke patients with upper extremity spasticity more than modified Ashworth scale ( MAS) 1+ and duration more than 6 months. Under different guidance methods (surface anatomy landmark/ ultrasonography /electric stimulation ), BTX-A will be injected to the key spastic muscles on upper extremity. Outcome measures include MAS, motor function ( Brunnstrom stage of upper extremity), range of motion , the degree and visual analog scale of pain , pinch and grasp power，Stroke Impact Scale, Barthel index and upper extremity function (Nine hole peg test，Action Reaearch Arm Test，Wolf Motor Function test，Chedoke Arm and Han Activity Inventory，Fugl-Meyer Assessment Scale，Motor Activity Log). All the assessments will be performed before BTX-A injection and followed up at 4 weeks, 8 weeks, 12 weeks and 24 weeks after injection. After performing all the assessments, investigators will investigate the efficiency of BTX-A by different guidance methods.

Four of arms:

ultrasonography direct-guidance: To inject Botulinum toxin type A on the spasticity lower extremity for stroke patients by Ultrasonography direct-guidance.

ultrasonography indirect-guidance: To inject Botulinum toxin type A on the spasticity lower extremity for stroke patients by Ultrasonography indirect-guidance.

electric stimulation guidance: To inject Botulinum toxin type A on the spasticity lower extremity for stroke patients by electric stimulation guidance.

surface anatomy landmark: To inject Botulinum toxin type A on the spasticity lower extremity for stroke patients by surface anatomy landmark.

ELIGIBILITY:
Inclusion Criteria:

* first onset.
* at least onset before 6 months.
* elbow, wrist and fingers are above Modified Ashworth Scale(MAS) 1+.
* Mini-Mental State Exam above 24.
* can follow all of the follow up and instruction.
* patients never accept botox, phenol and alcohol injections before.

Exclusion Criteria:

* contracture deformity on upper extremity.
* patients had accepted botox before or had have phenol, alcohol injections and operation 6 months ago.
* allergy to botox.
* have neither infection nor skin disorder on inject site.
* now accept aminoglycoside or other medicine treatment which may affect neuromuscular transition.
* combine other systemic disease of neurological or skelectomuscular system
* cognition disorder or aphasia after stroke.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-09; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth Scale | Change from Baseline Muscle Tone at 6 months
  patients will be evaluated at 4 weeks, 8 weeks, 12 weeks, 24 weeks after injection

SECONDARY OUTCOMES:
Brunnstrome Stage | Change from Baseline Condition at 6 months
  patients will be evaluated at 4 weeks, 8 weeks, 12 weeks, 24 weeks after injection
Active Range of Motion | Change from Baseline Data at 6 months
  patients will be evaluated at 4 weeks, 8 weeks, 12 weeks, 24 weeks after injection
4 Point Categorical Pain Intensity Scale | Change from Baseline Data at 6 months
  patients will be evaluated at 4 weeks, 8 weeks, 12 weeks, 24 weeks after injection
Hand-grasp strength Assessment | Change from Baseline Data at 6 months
  patients will be evaluated at 4 weeks, 8 weeks, 12 weeks, 24 weeks after injection
Pinch Strength Assessment | Change from Baseline Data at 6 months
  patients will be evaluated at 4 weeks, 8 weeks, 12 weeks, 24 weeks after injection
Barthel Index | Change from Baseline Data at 6 months
  patients will be evaluated at 4 weeks, 8 weeks, 12 weeks, 24 weeks after injection
Stroke Impact Scale (SIS) | Change from Baseline Data at 6 months
  patients will be evaluated at 4 weeks, 8 weeks, 12 weeks, 24 weeks after injection
Action Research Arm Test (ARAT) | Change from Baseline Data at 6 months
  patients will be evaluated at 4 weeks, 8 weeks, 12 weeks, 24 weeks after injection
Wolf Motor Function Test | Change from Baseline Data at 6 months
  patients will be evaluated at 4 weeks, 8 weeks, 12 weeks, 24 weeks after injection
Chedoke Arm and Hand Activity Inventory (CAHAI) | Change from Baseline Data at 6 months
  patients will be evaluated at 4 weeks, 8 weeks, 12 weeks, 24 weeks after injection
Fugl-Meyer Assessment | Change from Baseline Data at 6 months
  patients will be evaluated at 4 weeks, 8 weeks, 12 weeks, 24 weeks after injection
Motor Activity Log Scale | Change from Baseline Data at 6 months
  patients will be evaluated at 4 weeks, 8 weeks, 12 weeks, 24 weeks after injection
Nine Hole Peg Test | Change from Baseline Data at 6 months
  patients will be evaluated at 4 weeks, 8 weeks, 12 weeks, 24 weeks after injection

CONTACTS AND LOCATIONS:
Overall Officials: Pong Ya-Ping, MD, Study Chair — Rehabilitation
Locations (1):
- Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mizrahi EM, Angel RW. Impairment of voluntary movement by spasticity. Ann Neurol. 1979 Jun;5(6):594-5. doi: 10.1002/ana.410050620. No abstract available. PMID 475355
- [Background] Gracies JM, Nance P, Elovic E, McGuire J, Simpson DM. Traditional pharmacological treatments for spasticity. Part II: General and regional treatments. Muscle Nerve Suppl. 1997;6:S92-120. PMID 9826984
- [Background] Gracies JM, Elovic E, McGuire J, Simpson DM. Traditional pharmacological treatments for spasticity. Part I: Local treatments. Muscle Nerve Suppl. 1997;6:S61-91. PMID 9826983
- [Background] Difazio M, Jabbari B. A focused review of the use of botulinum toxins for low back pain. Clin J Pain. 2002 Nov-Dec;18(6 Suppl):S155-62. doi: 10.1097/00002508-200211001-00007. PMID 12569963
- [Background] Jankovic J. Botulinum toxin in clinical practice. J Neurol Neurosurg Psychiatry. 2004 Jul;75(7):951-7. doi: 10.1136/jnnp.2003.034702. PMID 15201348
- [Background] Lim EC, Seet RC. Use of botulinum toxin in the neurology clinic. Nat Rev Neurol. 2010 Nov;6(11):624-36. doi: 10.1038/nrneurol.2010.149. Epub 2010 Oct 12. PMID 21045798
- [Background] Brashear A, Gordon MF, Elovic E, Kassicieh VD, Marciniak C, Do M, Lee CH, Jenkins S, Turkel C; Botox Post-Stroke Spasticity Study Group. Intramuscular injection of botulinum toxin for the treatment of wrist and finger spasticity after a stroke. N Engl J Med. 2002 Aug 8;347(6):395-400. doi: 10.1056/NEJMoa011892. PMID 12167681
- [Background] Yablon SA, Brashear A, Gordon MF, Elovic EP, Turkel CC, Daggett S, Liu J, Brin MF. Formation of neutralizing antibodies in patients receiving botulinum toxin type A for treatment of poststroke spasticity: a pooled-data analysis of three clinical trials. Clin Ther. 2007 Apr;29(4):683-90. doi: 10.1016/j.clinthera.2007.04.015. PMID 17617291
- [Background] Yablon SA, Agana BT, Ivanhoe CB, Boake C. Botulinum toxin in severe upper extremity spasticity among patients with traumatic brain injury: an open-labeled trial. Neurology. 1996 Oct;47(4):939-44. doi: 10.1212/wnl.47.4.939. PMID 8857723
- [Background] Bakheit AM, Thilmann AF, Ward AB, Poewe W, Wissel J, Muller J, Benecke R, Collin C, Muller F, Ward CD, Neumann C. A randomized, double-blind, placebo-controlled, dose-ranging study to compare the efficacy and safety of three doses of botulinum toxin type A (Dysport) with placebo in upper limb spasticity after stroke. Stroke. 2000 Oct;31(10):2402-6. doi: 10.1161/01.str.31.10.2402. PMID 11022071
- [Background] Francisco GE. Botulinum toxin for post-stroke spastic hypertonia: a review of its efficacy and application in clinical practice. Ann Acad Med Singap. 2007 Jan;36(1):22-30. PMID 17285183
- [Background] Chin TY, Nattrass GR, Selber P, Graham HK. Accuracy of intramuscular injection of botulinum toxin A in juvenile cerebral palsy: a comparison between manual needle placement and placement guided by electrical stimulation. J Pediatr Orthop. 2005 May-Jun;25(3):286-91. doi: 10.1097/01.bpo.0000150819.72608.86. PMID 15832139
- [Background] Molloy FM, Shill HA, Kaelin-Lang A, Karp BI. Accuracy of muscle localization without EMG: implications for treatment of limb dystonia. Neurology. 2002 Mar 12;58(5):805-7. doi: 10.1212/wnl.58.5.805. PMID 11889247
- [Background] Lim EC, Ong BK, Seet RC. Botulinum toxin-A injections for spastic toe clawing. Parkinsonism Relat Disord. 2006 Jan;12(1):43-7. doi: 10.1016/j.parkreldis.2005.06.008. Epub 2005 Sep 29. PMID 16198612
- [Background] O'Brien CF. Injection techniques for botulinum toxin using electromyography and electrical stimulation. Muscle Nerve Suppl. 1997;6:S176-80. PMID 9826989
- [Background] Alter KE. High-frequency ultrasound guidance for neurotoxin injections. Phys Med Rehabil Clin N Am. 2010 Aug;21(3):607-30. doi: 10.1016/j.pmr.2010.05.001. PMID 20797552
- [Background] Berweck S, Schroeder AS, Fietzek UM, Heinen F. Sonography-guided injection of botulinum toxin in children with cerebral palsy. Lancet. 2004 Jan 17;363(9404):249-50. doi: 10.1016/S0140-6736(03)15351-2. No abstract available. PMID 14738817
- [Background] Schroeder AS, Berweck S, Lee SH, Heinen F. Botulinum toxin treatment of children with cerebral palsy - a short review of different injection techniques. Neurotox Res. 2006 Apr;9(2-3):189-96. doi: 10.1007/BF03033938. PMID 16785117
- [Background] Depedibi R, Unlu E, Cevikol A, Akkaya T, Cakci A, Cerekci R, Kose G, Unlusoy D. Ultrasound-guided botulinum toxin type A injection to the iliopsoas muscle in the management of children with cerebral palsy. NeuroRehabilitation. 2008;23(3):199-205. PMID 18560136
- [Background] Henzel MK, Munin MC, Niyonkuru C, Skidmore ER, Weber DJ, Zafonte RD. Comparison of surface and ultrasound localization to identify forearm flexor muscles for botulinum toxin injections. PM R. 2010 Jul;2(7):642-6. doi: 10.1016/j.pmrj.2010.05.002. PMID 20659720